CLINICAL TRIAL: NCT03120195
Title: EndoRotor® Ablation of Barrett's Esophagus: Safety and Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation for Liver Research (Other)
Collaborators: Interscope, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-688
Record Dates: First submitted 2017-04-04; First posted 2017-04-19 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Barretts Esophagus With Dysplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EndoRotor® ablation (Experimental): Prospective pilot study, to be performed in 30 patients with Barrett's esophagus that have an indication for ablation treatment. Barrett's ablation will be performed using the EndoRotor®.
  Interventions: Device: The EndoRotor®

INTERVENTIONS:
Device: The EndoRotor® — The EndoRotor® is in automated mechanical endoscopic mucosal resection system for use in the gastrointestinal tract. The EndoRotor suctions up the tissue and cuts it, automatically sending the tissue to a collection trap for histological evaluation.

SUMMARY:
The aim of this study is to assess the safety and feasibility of the EndoRotor® for the ablation of Barrett's esophagus.

DETAILED DESCRIPTION:
Prospective pilot study, to be performed in 30 patients with Barrett's esophagus that have an indication for ablation treatment. These include patients with low grade dysplasia (LGD), high grade dysplasia (HGD) or residual Barrett's after a complete endoscopic resection of a lesion containing HGD or esophageal adenocarcinoma. Ablation treatment will be performed by the EndoRotor ablation device, followed by surveillance endoscopy at 3 months where the feasibility for ablation will be assessed. During the 3 months follow-up, all adverse events such as perforation, post-procedural bleeding, stricture, and pain will be registered.

The EndoRotor® System is in automated mechanical endoscopic mucosal resection system for use in the gastrointestinal tract. The EndoRotor suctions up the tissue and cuts it, automatically sending the tissue to a collection trap for histological evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Age equal to or above 18 years (adult).
* Minimum (residual) Barrett's length of 2 cm and a maximum length of 5 cm (C0-5M2-5 according to the Prague classification)
* Scheduled Barrett's ablation for:

  * Histologically proven intestinal metaplasia with either high- or low-grade dysplasia in the absence of any visible lesion,
  * Residual Barrett's mucosa after complete endoscopic resection (for visible lesions containing HGD or EAC.) (EMR <50% of the circumference)
* Favorable anatomy (e.g. straight esophagus, no previous anti-reflux procedure) that allows performing endoscopic treatment with the EndoRotor®.

Exclusion Criteria:

* Presence of a visible lesion suspicious of early esophageal cancer or has a high chance of harboring cancer, or biopsy proven cancer.
* In case of previous EMR: EMR specimen showing deep submucosal invasion (> 500μm), poorly to undifferentiated cancer (G3 or G4), lymphovascular invasion, or positive vertical margins.
* In case of previous EMR: > 50% circumference.
* Any prior endoscopic ablation treatment or dilation for esophageal stenosis.
* Significant esophageal stenosis, preventing the passage of the therapeutic endoscope.
* Evidence of portal hypertension, esophageal varices, etc.
* An interval < 6 weeks between EMR and EndoRotor treatment.
* An interval of > 6 months after the last high resolution endoscopy with biopsies containing low or high grade dysplasia.
* Unable to undergo endoscopic procedure using sedation analgesics.
* Anti-coagulant therapy (apart from monotherapy aspirin) that cannot be discontinued prior to the procedure, OR uncorrectable hemostatic disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-01-27 (Actual); Primary Completion 2019-01-21 (Actual); Study Completion 2019-06-18 (Actual)

PRIMARY OUTCOMES:
Safety of EndoRotor® ablation of Barrett's mucosa; Number of participants with treatment related adverse events, such as bleeding, perforation or post procedural stenosis | 3 months
  Participants will have follow-up visits after the procedure during which the occurence of adverse events will be assessed. Adverse events will be classified according to the severity and onset timing.
Feasibility of EndoRotor® for the ablation of Barrett's mucosa | 3 months
  The percentage of endoscopically visible surface regression of Barrett's epithelium after 3 months post EndoRotor® treatment

SECONDARY OUTCOMES:
To assess the patient discomfort (recorded using the Numeric Rating Scale - grade 1-10) | 1 month
  The discomfort score will be recorded in a diary during the first 30 days post procedure
To assess the dysphagia-score (recorded using the Ogilvie score) | 1 month
  The dysphasia score will be recorded in a diary during the first 30 days post procedure
To assess a variety of symptoms (recorded using a 7 point Likert scale) | 1 month
  The symptoms will be recorded in a diary during the first 30 days post procedure
Total time to resect tissue | Procedure
  Procedure time is recorded during the EndoRotor® procedure
Ease of performing the EndoRotor® procedure | Procedure
  Procedural performance of the endoscopist will be assessed, using a predefined questionaire.

CONTACTS AND LOCATIONS:
Overall Officials: Arjun D. Koch, MD, PhD, Principal Investigator — Erasmus MC, University Medical Center Rotterdam
Locations (2):
- Netherlands (2):
  - Radboud University Medical Center, Nijmegen
  - Erasmus MC, University Medical Center, Rotterdam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gotink AW, Peters Y, Bruno MJ, Siersema PD, Koch AD. Nonthermal resection device for ablation of Barrett's esophagus: a feasibility and safety study. Endoscopy. 2022 Jun;54(6):545-552. doi: 10.1055/a-1644-4326. Epub 2021 Dec 21. PMID 34521118